CLINICAL TRIAL: NCT01244217
Title: An Open-label, Uncontrolled 4-week Study to Assess the Safety, Efficacy and Pharmacokinetics of Allegra® (Dry Syrup Formulation) 15 mg or 30 mg Twice Daily in Pediatric Patients With Perennial Allergic Rhinitis
Brief Title: Safety, Efficacy and Pharmacokinetic Study of Allegra in Pediatric Patients With Perennial Allergic Rhinitis (PAR)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SFY10717; U1111-1115-3842 (Other: UTN)
Record Dates: First submitted 2010-11-15; First posted 2010-11-19 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Rhinitis Perennial
MeSH Terms: interventions — fexofenadine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Age 6 months - 2 years (Experimental): Patients between 6 months and 2 years old
  Interventions: Drug: fexofenadine/Allegra (M016455)
- Age 2 - 11 years (Experimental): Patients between 2 and 11 years (and under 10.5 kg)
  Interventions: Drug: fexofenadine/Allegra (M016455)
- Age 2 - 11 years (and over 10.5 kg) (Experimental): Patients between 2 and 11 years (and over 10.5 kg)
  Interventions: Drug: fexofenadine/Allegra (M016455)

INTERVENTIONS:
Drug: fexofenadine/Allegra (M016455) — Pharmaceutical form:dry syrup formulation to be suspended in water
  Route of administration: oral

SUMMARY:
Primary Objective:

- To evaluate safety (4 weeks)

Secondary Objectives:

* To evaluate the long-term safety (12 weeks)
* To evaluate the efficacy
* To characterize the pharmacokinetic profile

DETAILED DESCRIPTION:
The study consists of four phases: up to 9-day screening phase, main 4-week treatment phase, up-to 8-week extension phase, and up-to 5-day post-treatment phase.

ELIGIBILITY:
Inclusion criteria:

* Aged 6 months through 11 years
* Patients with perennial allergic rhinitis

Exclusion criteria:

* Neither serum specific IgE antibody or skin reaction is positive for the antigen of perennial allergy.
* Nasal symptom score is 0 for either sneezing or nasal discharge, or sum of these two score is less than 3, or nasal congestion score is 4.
* Patients with vasomotor rhinitis or eosinophilic rhinitis.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 6 Months to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2010-10; Primary Completion 2011-07 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | 4 weeks
The number of clinically significant abnormalities for laboratory findings | 4 weeks

SECONDARY OUTCOMES:
Number of patients with adverse events | 12 weeks
The number of clinically significant abnormalities for laboratory findings | 12 weeks
Changes from baseline in nasal symptom scores on patient diary | 4 weeks
Changes from baseline in nasal symptom severity scores assessed by investigator or subinvestigator | week 2 and 4
Pharmacokinetic parameters of fexofenadine at steady state; AUC | week 4 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (15):
- Japan (15):
  - Sanofi-Aventis Investigational Site Number 392015, Fukuoka
  - Sanofi-Aventis Investigational Site Number 392012, Kanazawa
  - Sanofi-Aventis Investigational Site Number 392001, Kawaguchi-Shi
  - Sanofi-Aventis Investigational Site Number 392003, Kawasaki-Shi
  - Sanofi-Aventis Investigational Site Number 392004, Kawasaki-Shi
  - Sanofi-Aventis Investigational Site Number 392002, Kita-ku
  - Sanofi-Aventis Investigational Site Number 392011, Kofu
  - Sanofi-Aventis Investigational Site Number 392014, Obu-Shi
  - Sanofi-Aventis Investigational Site Number 392013, Seki-Shi
  - Sanofi-Aventis Investigational Site Number 392005, Yokohama
  - Sanofi-Aventis Investigational Site Number 392006, Yokohama
  - Sanofi-Aventis Investigational Site Number 392007, Yokohama
  - Sanofi-Aventis Investigational Site Number 392008, Yokohama
  - Sanofi-Aventis Investigational Site Number 392009, Yokohama
  - Sanofi-Aventis Investigational Site Number 392010, Yokohama